CLINICAL TRIAL: NCT04073511
Title: The Effectiveness and Safety of 'Eungyosan' and 'Samsoeum' for Common Cold - a Randomized, Parallel-group, Placebo-controlled, Multicenter Clinical Trial
Brief Title: Herbal Medicine 'Eungyosan' and 'Samsoeum' for Common Cold
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Principal Investigator, Jun-Yong Choi, Associate Professor, Korean Medicine Hospital of Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017012
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Common Cold
Keywords: Eungyosan; Samsoeum
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eungyosan (Experimental): Dosage is 1 packet, 2.3g, 3 times daily, 6.9g total daily dose. The total duration of administration is up to 8 days.
  Interventions: Drug: Eungyosan
- Samsoeum (Experimental): 3.37g of a packet, 3 times a day, the total daily dose is 10.11g. Total duration of administration is up to 8 days.
  Interventions: Drug: Samsoeum
- Placebo (Placebo Comparator): Take a total of 9.0g, 3.0g each, three times a day. The total duration of administration is up to 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eungyosan — This drug is a commercially available drug, manufactured according to the Preparation of granules, General rule of formulation, Korean Pharmacopoeia. Dosage is 1 packet, 2.3g, 3 times daily, 6.9g total daily dose. The total duration of administration is up to 8 days.
  Other Names: Hanpoong Eungyosan
  Arms: Eungyosan
Drug: Samsoeum — This drug is a commercially available drug, manufactured according to MFDS regulations and the Preparation of granules, General rule of formulation, Korean Pharmacopoeia. 3.37g of a packet, 3 times a day, the total daily dose is 10.11g. Total duration of administration is up to 8 days.
  Other Names: Hanpoong Samsoeum
  Arms: Samsoeum
Drug: Placebo — It is composed of lactose carb, corn starch, caramel pigment, and ginseng flavor powder. It is brown granule and made to be recognized as Korean medicine. Take a total of 9.0g, 3.0g each, three times a day. The total duration of administration is up to 8 days.
  Arms: Placebo

SUMMARY:
The investigators intend to conduct a multicenter clinical trial to verify the effectiveness and safety of the administration of 'Eungyosan(EGS)' and 'Samsoeum(SSE)' in cold patients.

DETAILED DESCRIPTION:
375 participants with symptoms of the common cold within 48 h will be recruited for this randomized, placebo-controlled trial. Subjects who will participate in the study will be divided into three groups, 'Eungyosan' group(EGS), 'Samsoeum' group(SSE) and placebo group according to the randomization number. Each group of subjects will take the drugs(EGS or SSE or placebo) 3 times a day up to 8 days.

The severity of illness will be assessed by Wisconsin Upper Respiratory Symptom Survey-21 Korean version (WURSS-21-K) and the VAS(visual analog scale) every 8days. Also, the duration of the common cold will be checked to evaluate the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged between 19 and 60 years as of the screening date
2. Onset of cold symptoms within 48 hours before screening
3. Those who have one or more of the symptoms and related symptoms of runny nose and sore throat (Related symptoms: nasal congestion, sneezing, sore throat, cough, sore throat, headache, chest tightness, fatigue)
4. Those who demonstrate understanding of the study details and have willingness to participate as evidenced by voluntary written informed consent
5. Those who can be followed up during the clinical trial
6. Those who do not meet the exclusion criteria

Exclusion Criteria:

1. Those who have sinusitis (when the sinus is opaque at the time of examination through the transillumination of the maxillary sinus and the frontal sinus), allergic rhinitis, pneumonia, flu (when coughing or sore throat with sudden fever above 38 ℃), bronchitis, otitis media, tonsillitis (PNS view, Chest Xray test if accurate test is needed)
2. Those who have chronic respiratory disease (chronic obstructive pulmonary disease, interstitial lung disease) and asthma
3. Those who have taken or should be taking or are taking antibiotics, antivirals, steroids, nasal decongestants, antihistamines, or other medications that are expected to alleviate cold symptoms, or those who have taken food that is expected to relieve cold symptoms within one week of the start of the study
4. Those who are being treated for liver cancer or cirrhosis, chronic renal failure, congestive heart failure, etc.
5. Those who have systemic disease or autoimmune disease which does not affect cold symptoms
6. Those who have severe mental illnesses such as depression or anxiety disorders, or those who are currently taking psychoneurological drugs such as antidepressants
7. Drug addicts or alcoholics
8. Alanine transaminase (ALT) or aspartate transaminase (AST) exceeds 3 times the upper limit of normal
9. Creatinine exceeds twice the upper limit of normal of the research institute
10. Weak person (less than body weight index (BMI) 18.5, clinically judged by Korean medical doctor through physical examination)
11. Those who have a weak stomach and are considered to be inadequate to take investigational drug (clinically judged by Korean medical doctor through physical examination)
12. Those who are with high blood pressure (vital sign measured at upper left after resting for at least 5 minutes at screening: systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥ 100 mmHg) or elderly
13. Those who have cardiac disorder or renal disorder (clinically judged by Korean medical doctor through physical examination, ECG, and serum biochemistry)
14. Those who have histories of hives, rash, or itching while taking medicines
15. Participants in other clinical trials within one month of the start of the trial (30 days prior to the screening visit) or plan to participate in other clinical trials during the trial
16. Pregnant women or women who may be pregnant
17. Those who do not agree to contraception in case of women of childbearing age
18. Those who are being held in group facilities such as social welfare facilities
19. Those who are inappropriate to participate in the trial by the investigator's judgment
20. Those who have hypersensitivity to the investigational drug (main ingredient and its components)
21. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
22. Those who have hypokalemia
23. Those who have difficulty in daily life due to sweats (excessive sweating, general weakness, etc.)
24. Those who have difficulty in daily life due to anorexia, nausea or vomiting
25. Those who are suspected of having pneumonia and need antibiotic treatment or those who are receiving medical treatment (those receiving other medications)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 375 (Estimated)
Dates: Start 2019-09-16 (Estimated); Primary Completion 2020-12-27 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The chance in total WURSS-21-K(Wisconsin Upper Respiratory Symptom Survey-21 Korean version) score | 6 days (Data collected at different times can be used as a reference)
  The investigators will assess the primary outcome through the change in total score(symptom score sum quality of life score) of Wisconsin Upper Respiratory Symptom Survey-21 Korean version (WURSS-21-K) 6 days after baseline. WURSS-21, which consists of questionnaires regarding gross severity, symptoms, quality of life, and improvement of illness. All items rank on a seven-point scale(1=very mild and 7=severe), where a higher score means higher severity. The symptom score is from 0(Do not have this symptom) to 70, and quality of life score is from 0(Not at all) to 56. Therefore, the total score ranges from 0 to 126.

SECONDARY OUTCOMES:
The change in WURSS-21-K(Wisconsin Upper Respiratory Symptom Survey-21 Korean version) symptom score | 6 days (Data collected at different times can be used as a reference)
  The investigators will assess the secondary outcome through the change in symptom score of Wisconsin Upper Respiratory Symptom Survey-21 Korean version (WURSS-21-K) 6 days after baseline. All items of symptom score rank on a seven-point scale(1=very mild and 7=severe), where a higher score means higher severity. The symptom score ranges from 0(Do not have this symptom) to 70.
The change in WURSS-21-K(Wisconsin Upper Respiratory Symptom Survey-21 Korean version quality of life score | 6 days (Data collected at different times can be used as a reference)
  The investigators will assess the secondary outcome through the change in quality of life score of Wisconsin Upper Respiratory Symptom Survey-21 Korean version (WURSS-21-K) 6 days after baseline. All items of quality of life score rank on a seven-point scale(1=very mildly and 7=severely), where a higher score means higher severity. The quality of life score ranges from 0(Not at all) to 56.
The duration of cold symptoms | up to 11 days
  The duration of cold symptoms
The change in the VAS(Visual Analogue Scale) | 6 days (Data collected at different times can be used as a reference)
  The investigators will assess the secondary outcome through the change in the VAS(Visual analog scale) 6 days after baseline, using EuroQol-visual analog scales(EQ-VAS). The EQ-VAS is a vertical visual analog scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which participants provide a global assessment of their health.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Yong Choi, PhD, Principal Investigator — Korean Medicine Hospital, Pusan National University
Locations (4):
- South Korea (4):
  - Korean Medicine Hospital, Pusan National University, Yangsan, Gyeongsangnam-do
  - Semyung University Korean Medicine Hospital, Jecheon, North Chungcheong
  - Korean Medicine Hospital of Daejeon University, Daejeon
  - KyungHee University Medical Center, Seoul

REFERENCES:
- [Derived] Kim KI, Hong M, Park YC, Lee BJ, Kim K, Kang BK, Choi JY. Effects of herbal medicines (Eunkyosan/Yin qiao san and Samsoeum/Shen su yin) for treating the common cold: A randomized, placebo-controlled, multicenter clinical trial. Integr Med Res. 2023 Dec;12(4):101005. doi: 10.1016/j.imr.2023.101005. Epub 2023 Oct 26. PMID 38033649
- [Derived] Kim KI, Hong M, Park YC, Lee BJ, Kim K, Kang BK, Choi JY. Herbal medicines (Eunkyosan and Samsoeum) for treating the common cold: a protocol for a randomized, placebo-controlled, multicenter clinical trial. Integr Med Res. 2020 Mar;9(1):48-53. doi: 10.1016/j.imr.2020.01.009. Epub 2020 Jan 22. PMID 32071868